CLINICAL TRIAL: NCT07133789
Title: The Contribution of Optical Mapping to the Characterization of Chromosomal Rearrangements in Patients With Neurodevelopmental Disorders
Acronym: Bionano
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP220309; IDRCB: 2022-A00020-43 (Registry Identifier: IDRCB ANSM)
Record Dates: First submitted 2025-06-23; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Anomalies Chromosome
MeSH Terms: conditions — Chromosome Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: blood sampling of all patients and their parents — blood sampling of all patients and their parents

SUMMARY:
In neurodevelomental disorders, duplications are genomic variations that are difficult to interpret because their orientation cannot be defined by conventional techniques (ACPA and FISH). However, their orientation determines whether a gene disruption and potential loss of function can be validated or not. The same applies to complex chromosomal rearrangements that can involve duplications and deletions, the interpretation of which is made difficult by the limitations of conventional techniques. The Bionano technique is an optical cartography genomic method that will provide access to this information by specifying both balanced and unbalanced chromosomal anomalies, their genomic location, and orientation. Our study is a prospective and multicentric (N=4) study involving 35 patients with neurodevelopmental disorders (NDD) and carrying a chromosomal anomaly identified by chromosomal microarray analysis (ACPA). Depending on the genetic anomaly, patients will be divided into two groups: patients carrying duplications containing or interrupting a gene already implicated in neurodevelopmental disorders. Duplications may involve the X chromosome and be present in male patients. The other group will involve NDD patients with a more complex chromosomal rearrangement (combination of deletion and duplication, ring chromosome structure, combination of multiple genomic imbalances). The optical genomic mapping (OGM) technology developed by Bionano Genomics is an innovative whole-genome exploration technology that enables the identification of balanced or unbalanced structural variants. OGM is based on specific labeling of repetitive regions following extraction of high molecular weight DNA (fragments ranging from 100kb to 2Mb). The algorithms associated with this new technology allow the identification of balanced structural rearrangements as small as 500bp and unbalanced rearrangements as small as 5kb. This technique also enables the physical localization of each analyzed region, characterizing insertions, deletions, duplications, repeat expansions, inversions, and translocations.

Finally, in the first group, this technology is expected to allow us to characterize the breakpoints and orientation of duplicated segments in order to better understand the functional impact on the interrupted gene. Indeed, duplication can result in obtaining a complete additional copy of the gene, disrupt the gene leading to its misregulation (equivalent to a loss-of-function variation), disrupt another gene if the duplicated segment is inserted elsewhere in the genome or if it involves a regulatory region, or have no effect on gene expression. Similarly, in the second group, this technique will allow us to characterize the complex chromosomal rearrangement at the molecular level and define its functional impact.

This technology will enable us to better understand the pathophysiology of pediatric neurodevelopmental disorders (NDD) and guide the genetic counseling provided to the patient and their family. Furthermore, more generally, the results will help us better understand the complex architecture of neurodevelopmental disorders, ultimately allowing for more targeted therapeutic solutions. Finally, our study will assess the contribution of this technique and its feasibility in routine clinical practice.

DETAILED DESCRIPTION:
Neurodevelopmental disorders (NDD) affect almost 10% of the general population, and encompass a very broad spectrum of manifestations linked to an abnormality in brain development. They include intellectual disability (ID), autism spectrum disorders (ASD), pervasive developmental disorders (PDD), epilepsy or even DYS disorders (dyslexia, dyspraxia...) or attention deficit disorder with or without hyperactivity (ADHD) (Thapar, Cooper, & Rutter, 2017). These signs appear early, usually in childhood, and can progress into adulthood. Moreover, these disorders are frequently associated with each other and present with degrees of severity that vary widely from one patient to another. The genetic architecture of TND is complex, and remains poorly understood in some cases, despite the advent of new diagnostic technologies in human genetics. Currently, first-line genetic explorations, chromosomal analysis by microarray (ACPA) and high throughout sequencing enable a diagnosis to be made in 15-20% and 25-35% of cases respectively (Martin & Ledbetter, 2017; Vasudevan & Suri, 2017).

The interpretation of CNVs depends on many well-established parameters such as the nature of the variation (deletions are often more penetrant than duplications), size, gene content and heritability (Riggs et al.). Some recurrent CNVs are associated with specific phenotypes and their interpretation is unambiguous. Other non-recurrent CNVs are more difficult to interpret, particularly duplications, since they concern genes involved in NDD, or in essential developmental functions, notably brain development. The functional impact of duplications depends on their location, orientation (tandem or inverted) and whether or not an intact copy of the gene of interest is maintained. A whole-genome sequencing (WGS) study of 184 patients with duplications showed that in the majority of cases (83%), the duplicated segment was oriented in tandem and therefore had no functional consequences, and that in 2.8% of cases, this segment (inverted or inserted elsewhere) was at the origin of the gene dysregulation mechanism involved in the abnormal phenotype (Newman et al.). More complex chromosomal rearrangements, such as chromothripsis, complex translocations or atypical chromosomal rearrangements, are sometimes revealed by ACPA or exome sequencing techniques, but the mechanisms of occurrence escape these classic technologies.Optical genomic mapping (OGM) developed by Bionano Genomics is an innovative genome-wide scanning technology that enables the identification of balanced or unbalanced structural variants in diagnosis, as described in studies by Bocklandt et al. and more recently by the team of Mantere et al. Optical mapping is based on specific marking of repeated regions after extraction of high molecular weight DNA (100kb to 2Mb fragments). The algorithms associated with this new technology enable the identification of balanced structural rearrangements as early as 500bp, and unbalanced rearrangements as early as 5kb. This technique also enables the physical localization of each analyzed region, characterizing insertions, deletions, duplications, repeat expansions, inversions and translocations (Chan et al.).

This technology should enable us to characterize the breakpoints and orientation of duplicated segments to better understand the functional impact on the interrupted gene. Duplication can induce an additional complete copy of the gene, disrupt the gene leading to its misregulation (equivalent to a loss-of-function variation), disrupt another gene if the duplicated segment is inserted elsewhere in the genome or if it concerns a regulatory region, or have no effect on gene expression.

Hypothesis of the study and objectives :

In patients with TND, some CNVs are considered as variants of unknown significance (VOUS)"" when the classification criteria do not allow us to decide whether or not they are pathogenic; particularly, duplications involving genes of interest in neurodevelopment, where the impact on gene expression is uncertain. Qualitative knowledge of the structure of these anomalies, such as the direction of duplication or the position of insertion in the genome, could enable us to understand the effect on gene expression.

OGM technology provides access to this qualitative information, allowing us to make a genetic diagnosis in these patients: i/A tandem duplication would have no impact on gene expression, leaving two intact copies of the gene; ii/Inversion of the duplicated segment could result in loss of function of the gene; iii/insertion of the duplicated segment at another locus could deregulate the interest gene but also could modify the expression of other genes.

In cases of complex rearrangements identified by ACPA, qualitative data from OGM can help to understand the chromosomal mechanisms. Precise knowledge of these mechanisms can drive appropriate genetic counseling, particularly when the duplication is located on the X chromosome and transmitted by the mother of the affected child.

In addition, the higher resolution of OGM compared with ACPA could revealed other CNVs that also could be implicated in the abnormal phenotype.

Studied population and experimental scheme :

Our prospective multicentric (4 centers in Robert Debré hospital) study will include 35 patients with NDD and a chromosomal abnormality identified in ACPA. Depending on the genetic abnormality, patients were distributed in two groups:

Around half the patients carried duplications involving or interrupting a gene already implicated in NDD. Duplications may involve the X chromosome and be present in male patients. In the other group, half of the patients presented with a more complex chromosomal rearrangement (combination of deletion and duplication, ring chromosome structure, combination of several genomic imbalances).

Both parents will also be sampled and will be considered as ""controls"" for the study.

After informations gived to the family during a follow-up visit, an inclusion visit after 15 days will collect the necessary consent and peripheric blood samples of the patient and his parents.

Samples are sent to the Institut Curie (Genomics Platform - Department of Translational Research). The analytical phase is carried out at the Institut Curie: high molecular weight DNA extraction and Bionano technique. Data are transmitted to Robert Debré's cytogeneticists, who interpret the results.

The patients will be included for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients: children aged 2 and over at the time of inclusion (and up to 20 years of age)
* Patients followed at Robert Debré for TND who, as part of their care,
* who have undergone chromosomal analysis by DNA microarray (ACPA) which has identified a chromosomal abnormality of difficult interpretation (duplication or complex rearrangement).

Exclusion Criteria:

* Patients without medical insurance

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Both parents of each patient will also be sampled to facilitate interpretation of the genomic data and to clarify the segregation of chromosomal rearrangements identified in their child. In the case of chromosomal abnormalities on the X chromosome in a boy, the absence of the father will not be limiting.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2022-07-12 (Actual); Primary Completion 2024-07-12 (Actual); Study Completion 2025-08-19 (Estimated)

PRIMARY OUTCOMES:
Precise characterization of chromosomal segments involved in duplications or complex chromosomal rearrangements identified in ACPA | 24 months
  chromosomal segments involved in duplications or complex chromosomal rearrangements identified in ACPA are characterized by:
  * the size in kb
  * the orientation
  * the genomic position

CONTACTS AND LOCATIONS:
Locations (1):
- Robert Debré Hospital, Paris, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided